CLINICAL TRIAL: NCT05883254
Title: Detection of RNA Binding Protein Pumilio1 (PUM1) Expression in Patients With Sickle Cell Anemia and β-thalassemia Intermedia
Brief Title: Pumilio1 (PUM1) Expression, Sickle Cell Anemia, β-thalassemia Intermedia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mervat Awad Mohamed Ibrahim, asssistant lecturer, Assiut University
Other Study IDs: PUM1 Sickle cell Thalassemia
Record Dates: First submitted 2023-05-21; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Sickle Cell Disease, Beta Thalassemia Intermedia
MeSH Terms: conditions — Anemia, Sickle Cell; beta-Thalassemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Normal individuals
  Interventions: Diagnostic Test: RNA Binding Protein Pumilio1 (PUM1) Expression by reverse transcriptase quantatative PCR
- thalassemia intermedia patients and sickle cell disease patients: 1. Inclusion criteria
     * Patients with sickle cell anemia and β-thalassemia intermedia.
     * Patients are of both sexes (males and females) at any age.
  2. Exclusion criteria:
     * Patients with any other type of haemolytic anaemias.
     * Patients on Hydroxyurea therapy.
  Interventions: Diagnostic Test: RNA Binding Protein Pumilio1 (PUM1) Expression by reverse transcriptase quantatative PCR

INTERVENTIONS:
Diagnostic Test: RNA Binding Protein Pumilio1 (PUM1) Expression by reverse transcriptase quantatative PCR — Quantatative Real -Time PCR for quantification of PUM1;
  * The type of the recruited samples: Ethylenediamine tetra-acetic acid (EDTA) peripheral blood samples.
  * The method of total RNA extraction: TRIzol and TRIzol LS.
  * The purity and concentration of the RNA were measured using a Nano Drop 2000 instrument.
  * cDNA was amplified with primers using the GoScript Reverse Transcription system.
  Western Blotting Assay of PUM1 protein levels
  Other Names: Western Blotting Assay of PUM1 protein levels

SUMMARY:
1. To study the expression pattern of PUM1 gene in patients with sickle cell anemia and β-thalassemia intermedia.
2. To detect PUM1 protein levels in sickle cell anemia and β-thalassemia intermedia patients.
3. To correlate PUM1 gene expression pattern and protein levels with HbF levels in sickle cell anemia and β-thalassemia intermedia patients.

DETAILED DESCRIPTION:
The disorders of β-hemoglobin, sickle cell disease (SCD) and β-thalassemia, are major causes of morbidity and mortality worldwide. These diseases are the most common genetic disorders in the world.

SCD is due to a single base-pair point mutation in the β-globin gene resulting in the substitution of valine for glutamic acid in the β-globin chain. The pathophysiology is directly related to polymerization of deoxygenated hemoglobin, leading to a cascade of pathologic events including erythrocyte sickling, vaso-occlusion, and hemolysis.

In β-thalassemia, insufficient production of the β-globin molecule results in an excess of free α-globin chains that can precipitate within erythroid precursors, impairing their maturation and leads to death of these precursors and ineffective production of erythroid cells. As a result, a significant anemia occurs and the consequent expansion of erythroid precursors can lead to secondary problems in bones and other organs.

The hemoglobin molecule is a tetramer composed of two subunits of α-like globin peptides and two subunits of the β-like globin peptides, along with heme moieties. β-globin switching from fetal γ-globin (HBG1 and HBG2) to adult β-globin is a developmental process that occurs in erythrocytes at around the time of birth. Fetal hemoglobin (HbF) induction in adult erythrocytes is an effective therapeutic strategy for SCD and β-thalassemia.

Pumilio1 (PUM1) is a novel target of the erythroid master transcription factor erythroid Krüppel-like factor (EKLF). PUM1 is a member of Pumilio-Fem3-binding factor (PUF) family of sequence specific RNA-binding proteins, acts as a posttranscriptional repressor by binding to the 3' untranslated region (3'-UTR) of messenger RNA (mRNA). It peaks during terminal erythroid differentiation and binds to fetal γ-globin (HBG1) mRNA and impairs its stability and translation. HBG1 has 2 core PUM1 consensus binding sites, but HBG2 and adult globins do not. Knockdown of PUM1 leads to a robust increase in HBF (∼22%) without affecting β-globin levels in human erythroid cells. Moreover, targeting PUM1 does not affect erythropoiesis, which provides a potentially safe and effective therapeutic strategy for SCD and β-thalassemia. Also it was found that elevated HbF levels in the absence of anemia in an individual with a novel heterozygous PUM1 mutation in the RNA-binding domain, which suggests that PUM1 is a critical player during human hemoglobin switching.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sickle cell anemia and β-thalassemia intermedia.
* Patients are of both sexes (males and females) at any age.

Exclusion Criteria:

* Patients with any other type of haemolytic anaemias.
* Patients on Hydroxyurea therapy.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with sickle cell anemia and β-thalassemia intermedia
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Expression pattern of PUM1 gene in patients with sickle cell anemia and β-thalassemia intermedia. | saple taken after diagnosis and before recieve treatment. If patients already on treatment , sample taken at least one month after stoppage of hydroxyurea or blood transfusion
  Detect PUM1 protein levels in sickle cell anemia and β-thalassemia intermedia patients and to correlate PUM1 gene expression pattern and protein levels with HbF levels in sickle cell anemia and β-thalassemia intermedia patients.

REFERENCES:
- [Background] Persons DA. Hematopoietic stem cell gene transfer for the treatment of hemoglobin disorders. Hematology Am Soc Hematol Educ Program. 2009:690-7. doi: 10.1182/asheducation-2009.1.690. PMID 20008255
- [Background] Sankaran VG, Orkin SH. The switch from fetal to adult hemoglobin. Cold Spring Harb Perspect Med. 2013 Jan 1;3(1):a011643. doi: 10.1101/cshperspect.a011643. PMID 23209159
- [Background] Sankaran VG, Nathan DG. Reversing the hemoglobin switch. N Engl J Med. 2010 Dec 2;363(23):2258-60. doi: 10.1056/NEJMcibr1010767. No abstract available. PMID 21121839
- [Background] Nuinoon M, Makarasara W, Mushiroda T, Setianingsih I, Wahidiyat PA, Sripichai O, Kumasaka N, Takahashi A, Svasti S, Munkongdee T, Mahasirimongkol S, Peerapittayamongkol C, Viprakasit V, Kamatani N, Winichagoon P, Kubo M, Nakamura Y, Fucharoen S. A genome-wide association identified the common genetic variants influence disease severity in beta0-thalassemia/hemoglobin E. Hum Genet. 2010 Mar;127(3):303-14. doi: 10.1007/s00439-009-0770-2. PMID 20183929
- [Background] Stamatoyannopoulos G. Control of globin gene expression during development and erythroid differentiation. Exp Hematol. 2005 Mar;33(3):259-71. doi: 10.1016/j.exphem.2004.11.007. PMID 15730849
- [Background] Elagooz R, Dhara AR, Gott RM, Adams SE, White RA, Ghosh A, Ganguly S, Man Y, Owusu-Ansah A, Mian OY, Gurkan UA, Komar AA, Ramamoorthy M, Gnanapragasam MN. PUM1 mediates the posttranscriptional regulation of human fetal hemoglobin. Blood Adv. 2022 Dec 13;6(23):6016-6022. doi: 10.1182/bloodadvances.2021006730. PMID 35667093
- [Background] Goldstrohm AC, Hall TMT, McKenney KM. Post-transcriptional Regulatory Functions of Mammalian Pumilio Proteins. Trends Genet. 2018 Dec;34(12):972-990. doi: 10.1016/j.tig.2018.09.006. Epub 2018 Oct 10. PMID 30316580